CLINICAL TRIAL: NCT07012642
Title: Efficacy of GLP-1 Receptor Agonists in Treating Upper and Lower Extremity Lymphedema
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Advanced Reconstructive Surgery Alliance (Other Government)
Responsible Party: Principal Investigator, Joseph Dayan, Principal Investigator, Advanced Reconstructive Surgery Alliance
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLP-1 in Lymphedema
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lymphedema
Keywords: Efficacy of GLP-1 in lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Experimental): Participants will received GLP-1 RAs for 6 months to study the effects on lymphedema.
  Interventions: Drug: GLP-1 Receptor Agonists

INTERVENTIONS:
Drug: GLP-1 Receptor Agonists — GLP-1 RAs in lymphedema

SUMMARY:
Lymphedema affects millions and currently lacks effective drug treatments, relying mainly on compression therapy. Glucagon-like peptide-1 receptor agonists (GLP-1 RAs) have shown potential in managing obesity and diabetes, which can worsen lymphedema. Although anecdotal evidence suggests benefits of GLP-1 RAs for lymphedema patients, rigorous prospective studies are lacking. This study aims to evaluate the effectiveness of GLP-1 RAs in improving quality of life and clinical outcomes in lymphedema patients, thereby addressing a critical gap in literature and potentially offering a new treatment option.

DETAILED DESCRIPTION:
Research Protocol: GLP-1Ras - Investigator-Initiated Study

Principal Investigator: Joseph Dayan, MD, MBA

Title: Efficacy of GLP-1 Receptor Agonists in Treating Upper and Lower Extremity Lymphedema

Background and Rationale

Introduction: Lymphedema is an incurable and relentless progressive disease marked by swelling of the upper or lower limb requiring life-long compression. Patients have a high risk of cellulitis and deteriorating quality of life. Lymphedema is a major public health problem with an estimated incidence in the United States of 5 million. There is no cure and no drug to treat this disease.

Literature Review: Glucagon-like peptide-1 receptor agonists (GLP-1 RAs) are now ubiquitous in the United States given their effectiveness in treating obesity and diabetes. Elevated BMI and insulin resistance have been widely reported to worsen lymphedema. Consequently, GLP-1 RAs may have a positive effect on lymphedema. Anecdotally we have observed patients with chronic lymphedema dramatically improve after taking GLP-1 receptor agonists but there is currently no prospective data available.

Rationale: Lymphedema affects millions and currently lacks effective drug treatments, relying mainly on compression therapy. Glucagon-like peptide-1 receptor agonists (GLP-1 RAs) have shown potential in managing obesity and diabetes, which can worsen lymphedema. Although anecdotal evidence suggests benefits of GLP-1 RAs for lymphedema patients, rigorous prospective studies are lacking. This study aims to evaluate the effectiveness of GLP-1 RAs in improving quality of life and clinical outcomes in lymphedema patients, thereby addressing a critical gap in literature and potentially offering a new treatment option.

Objectives

Primary Objective: To evaluate the quality-of-life improvements following GLP-1 RA treatment, utilizing the Lymphedema Life Impact Scale (LLIS) as a measurement tool.

Secondary Objectives: To evaluate the efficacy of GLP-1 RAs in reducing limb volume, bioimpedance, compression use, and incidence of cellulitis.

Hypotheses

GLP-1 receptor agonists will improve quality of life and reduce limb volume in lymphedema patients.

Study Design

Type of Study: Prospective, Single arm study, off-label use of GLP-1 receptor agonists to treat upper or lower extremity lymphedema.

Duration: 24 Months

Study Setting: Conduct at an outpatient lymphedema clinic

Population: Adults with Upper and lower extremity Lymphedema, (ISL) stages II and II

Sample Size: 110 participants

Follow-up Visits: Baseline, 3 months, and 6 months post-treatment visit

Participants

Eligibility Criteria

Inclusion Criteria:

Adults 18 years or older with unilateral upper or lower extremity lymphedema Limb volume > 5% BMI => 23 Oncology clearance if there is a cancer history

Exclusion Criteria:

Moderate to severe venous insufficiency Actively using GLP-1 RAs Known intolerance or adverse effect to GLP-1 RAs Medical history or morbidity where GLP-1 RAs are contraindicated as per patient's primary care provider such as MEN syndrome or history of thyroid cancer

Methods

Data Collection:

Lymphedema Life Impact Scale score (validated patient-reported outcome metric) Limb volume Bioimpedance BMI Compression use Incidence of cellulitis

Interventions: GLP-1 RA treatment will be administered by the patient's primary provider for 6 months.

Outcome Measures

Primary Outcome:

Patient reported quality of life outcome (Lymphedema Life Impact Scale)

Secondary Outcomes:

Limb volume Bioimpedance BMI Incidence of cellulitis Compression use

Data Analysis Plan

Statistical Methods:

Utilize appropriate statistical tests, including a t-test with an effect size of 0.15 and a power of 0.95.

To adequately power this study, 74 participants are needed to complete a 6-month course of GLP-1 RA treatment and follow-up. Assuming a dropout rate of 30%, we plan to enroll 110 patients to meet this goal.

Software:

IBM SPSS for data analysis.

Handling Missing Data:

To address missing data, all instances will be documented, and efforts will be made to recover missing information. Multiple imputation techniques will be used to estimate missing values for continuous variables, such as limb volume and LLIS scores. Sensitivity analyses will be conducted to evaluate the impact of missing data on study outcomes, ensuring robustness and transparency in the study's findings.

Ethical Considerations

Informed Consent:

Participants will provide informed consent, understanding the study's scope and procedures.

Confidentiality:

Participant data will be kept confidential, adhering to ethical standards.

Approval:

Ethical approval will be obtained from a relevant ethics committee or institutional review board (IRB).

Study Timeline Estimated Start Date: April 9, 2025

Estimated Completion Date: April 9, 2027

Recruitment:

Recruit patients from internal lymphedema population Clinicaltrials.gov Patient referrals from other providers and social media

Budget and Funding

Budget:

No anticipated study costs. The study participation is voluntary

Funding Sources:

The project is currently not funded

Potential Risks and Benefits

Risks, benefits, and alternatives to GLP-1 RA treatment will be discussed with the patient in addition to the patient reviewing this consideration with their provider.

The most common adverse event from GLP-1 treatment is gastrointestinal intolerance such as nausea or vomiting (5% incidence).

Adverse events:

The site will begin to report AE/SAE after the patient signs the informed consent.

All serious adverse events (SAEs) will be documented and reported to the Institutional Review Board (IRB) within 24 hours of the patient site becoming aware.

Participant Discontinuation/ Withdrawal from the study:

Participants have the right to withdraw from the study at any time upon their request.

Dissemination Plan:

The results of the study will be submitted as a research manuscript for publication in a peer-reviewed journal either the New England Journal of Medicine or the Journal of the American Medical Association.

ELIGIBILITY:
Inclusion Criteria:

Adults 18 years or older with unilateral upper or lower extremity lymphedema Limb volume > 5% BMI => 23 Oncology clearance if there is a cancer history

Exclusion Criteria:

Moderate to severe venous insufficiency Actively using GLP-1 RAs Known intolerance or adverse effect to GLP-1 RAs Medical history or morbidity where GLP-1 RAs are contraindicated as per patient's primary care provider such as MEN syndrome or history of thyroid cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-04-09 (Estimated); Study Completion 2027-04-09 (Estimated)

PRIMARY OUTCOMES:
Patient reported quality of life outcome using LLIS | 6 months
  Lymphedema Life Impact Scale

SECONDARY OUTCOMES:
Physiological improvement | 6 months
  Limb volume Bioimpedance BMI Incidence of cellulitis Compression use

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - River Center, Red Bank, New Jersey
  - 260 Old Hook Rd Suite 304, Westwood, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
De-identified study results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the conclusion of the study (start date) For five years (end date)
Access Criteria: All de-identified study documents will be available.